CLINICAL TRIAL: NCT02874014
Title: Prospective Evaluation of Hypofractionation Proton Beam Therapy With Concurrent Treatment of the Prostate and Pelvic Nodes for Clinically Localized, High Risk or Unfavorable Intermediate Risk Prostate Cancer
Brief Title: Hypofractionation Proton Beam Therapy With Concurrent Treatment of Prostate and Pelvic Nodes for Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1651; MC1651 (Other: Mayo Clinic); 15-009528 (Other: Mayo Clinic Institutional Review Board); NCI-2017-02364 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2016-08-17; First posted 2016-08-22 (Estimated); Results first posted 2023-07-10 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-07

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hypofractionation Proton beam therapy (Experimental): Hypofractionation Proton beam therapy with Concurrent Treatment of the Prostate and Pelvic Nodes
  Interventions: Radiation: Hypofractionation Proton beam therapy with Concurrent Treatment of the Prostate and Pelvic Nodes

INTERVENTIONS:
Radiation: Hypofractionation Proton beam therapy with Concurrent Treatment of the Prostate and Pelvic Nodes

SUMMARY:
The study is to examine a moderate hypofractionation regimen of proton beam therapy for high risk or unfavorable intermediate risk prostate cancer. The prostate and seminal vesicles are treated with 6750 centigray (RBE) in 25 fractions (i.e. 270 centigray/fraction), while the regional pelvic nodes receive 4500 centigray (RBE) in 25 fractions (i.e. 180 centigray/fraction) simultaneously. The overall treatment time is 5 weeks.

DETAILED DESCRIPTION:
Proton beam therapy can provide a therapeutic gain by offering at least equivalent (or superior) tumor control while reducing the risk of radiation toxicity, in comparison with conventional photon-based external beam radiotherapy, given its dose-deposition characteristics. Currently the clinical target volume of proton beam for the treatment of prostate cancer has been mostly limited to the prostate and the seminal vesicles. There has been no study of proton beam therapy to treat both the primary tumor in the prostate and the regional pelvic nodes simultaneously using a moderate hypofractionation regimen.

The study is a prospective, single-arm, clinical trial to evaluate a moderate hypofractionation regimen of proton beam therapy for high risk or unfavorable intermediate risk prostate cancer. The clinical target volumes of proton beam therapy include both the prostate/seminal vesicles and the regional pelvic nodes. The primary objective is to assess late grade ≥ 3 gastrointestinal (GI) and genitourinary (GU) toxicity. The secondary objectives are to evaluate late grade ≥ 2 GI and GU toxicity, acute grade ≥ 3 GI and GU toxicity, and disease-free survival including freedom from PSA (prostate specific antigen) relapse at 5 years. The study provides an avenue to examine the safety, efficacy, cost effectiveness, and convenience of a moderate hypofractionation regimen (5-week course) of proton beam therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male; Age ≥ 18 years.
* Histological confirmation of adenocarcinoma of the prostate within 6 months of study enrollment.
* Clinical stage T1-2 N0 M0, Gleason Score 7, Prostate Specific Antigen (PSA) 20-100 ng/mL, or Clinical stage Any T N0 M0, Gleason Score 8-10, PSA ≤ 100 ng/mL, or Clinical stage T3-4 N0 M0, any Gleason Score, PSA ≤ 100 ng/mL, or Clinical stage T1-2 N0 M0, Gleason Score 4+3, PSA 10-20 ng/mL
* Zubrod performance score (PS) ≤ 1
* Total bilirubin, aspartate aminotransferase, alkaline phosphatase, and serum creatinine: < 2 x upper normal limit
* Signed informed consent.

Exclusion Criteria:

* Any known nodal (N1) or distant metastasis (M1)
* Previous androgen deprivation therapy lasting more than 6 months
* History of inflammatory bowel disease
* Presence of a hip prosthesis
* Prior pelvic radiotherapy or prostatectomy
* Prior or concurrent antineoplastic agents (chemotherapy)
* Previous or concurrent malignancy other than non-melanoma skin cancer within 5 years of diagnosis of prostate cancer.
* Inability to start the protocol treatment within 1 month after study enrollment.
* Medical or psychiatric conditions that preclude informed decision-making or compliance with the protocol treatment or follow-up

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2016-07-25 (Actual); Primary Completion 2021-02-08 (Actual); Study Completion 2025-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark R. Waddle, MD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- [Derived] Choo R, Hillman DW, Mitchell C, Daniels T, Vargas C, Rwigema JC, Corbin K, Keole S, Vora S, Merrell K, Stish B, Pisansky TM, Davis BJ, Amundson A, Wong W. Five-Year Outcomes of Moderately Hypofractionated Proton Therapy Incorporating Elective Pelvic Nodal Irradiation for High-Risk Prostate Cancer. Int J Radiat Oncol Biol Phys. 2025 May 1;122(1):99-108. doi: 10.1016/j.ijrobp.2024.11.115. Epub 2024 Dec 11. PMID 39672515
- [Derived] Choo R, Hillman DW, Mitchell C, Daniels T, Vargas C, Rwigema JC, Corbin K, Keole S, Vora S, Merrell K, Stish B, Pisansky T, Davis BJ, Amundson A, Wong W. Late Toxicity of Moderately Hypofractionated Intensity-Modulated Proton Therapy Treating the Prostate and Pelvic Lymph Nodes for High-Risk Prostate Cancer. Int J Radiat Oncol Biol Phys. 2023 Apr 1;115(5):1085-1094. doi: 10.1016/j.ijrobp.2022.11.027. Epub 2022 Nov 22. PMID 36427645
- [Derived] Choo R, Hillman DW, Daniels T, Vargas C, Rwigema JC, Corbin K, Keole S, Vora S, Merrell K, Stish B, Pisansky T, Davis B, Amundson A, Wong W. Proton Therapy of Prostate and Pelvic Lymph Nodes for High Risk Prostate Cancer: Acute Toxicity. Int J Part Ther. 2021 Sep 14;8(2):41-50. doi: 10.14338/IJPT-20-00094.1. eCollection 2021 Fall. PMID 34722810
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Hypofractionation Proton Beam Therapy: Hypofractionation Proton beam therapy with Concurrent Treatment of the Prostate and Pelvic Nodes>>>
  >>>>
  >>>
  >>>> Hypofractionation Proton beam therapy with Concurrent Treatment of the Prostate and Pelvic Nodes
Period: Overall Study
Arm/Group | Hypofractionation Proton Beam Therapy
Started | 56
Completed | 54
Not Completed | 2

BASELINE CHARACTERISTICS:
Groups:
- Hypofractionation Proton Beam Therapy: Hypofractionation Proton beam therapy with Concurrent Treatment of the Prostate and Pelvic Nodes>>>>
  >>>> Hypofractionation Proton beam therapy with Concurrent Treatment of the Prostate and Pelvic Nodes
Arm/Group | Hypofractionation Proton Beam Therapy
Number analyzed (Participants) | 54
Age, Continuous [Median (Full Range); unit: years] | 75.5 [55 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 51
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 0
  White | 49
  More than one race | 0
  Unknown or Not Reported | 3
Performance status (ECOG) [Count of Participants; unit: Participants] — 0: Asymptomatic and fully active.>>>
  1: Symptomatic; fully ambulatory; restricted in physically strenuous activity.>>> ECOG = 0 is better. ECOG = 1 is worse.
  Participants
    ECOG score 0 | 47
    ECOG score 1 | 7
BMI [Median (Full Range); unit: kg/m^2] | 29.0 [21.9 to 35.0]
Prostate volume (mL) [Median (Inter-Quartile Range); unit: mL] | 41.1 [32.3 to 54.7]
History of prior TURP [Count of Participants; unit: Participants]
  Yes | 5
  No | 49
Use of alpha-1 blocker [Count of Participants; unit: Participants]
  Yes | 5
  No | 49
Use of antiplatelet or anticoagulant medication [Count of Participants; unit: Participants]
  Yes | 11
  No | 43
Baseline IPSS score [Count of Participants; unit: Participants] — A score of 0 to 7 indicates mild symptoms, 8 to 19 indicates moderate symptoms and 20 to 35 indicates severe symptoms Population: Two patients are missing scores
  Participants
    0-7: number analyzed (Participants) | 52
    0-7 | 28
    8-19: number analyzed (Participants) | 52
    8-19 | 22
    20-35: number analyzed (Participants) | 52
    20-35 | 2
Gleason score [Count of Participants; unit: Participants] — The Gleason score usually ranges from 6 to 10. The lower the Gleason score, the more the cancer cells look like normal cells and are likely to grow and spread slowly.
  Participants
    6 | 4
    7 | 17
    8-10 | 33
Baseline PSA, ng/mL [Median (Full Range); unit: ng/mL] | 10.7 [0.65 to 97.3]
T stage [Count of Participants; unit: Participants] — T1 means the cancer is too small to be seen on a scan, or felt during an examination of the prostate. T2 means the cancer is completely inside the prostate gland. T3a means the cancer has broken through the capsule (covering) of the prostate gland. T3b means the cancer has spread into the tubes that carry semen (seminal vesicles). T4 means the cancer has spread into other body organs nearby, such as the back passage, bladder, or the pelvic wall.
  Participants
    T1-T2 | 23
    T3a | 21
    T3b | 10
    T4 | 0
Risk [Count of Participants; unit: Participants]
  High-risk | 52
  Unfavorable intermediate risk | 2
Duration of ADT (mo) [Median (Full Range); unit: months] | 18.1 [4.0 to 36.8]

OUTCOME MEASURES:

1. Primary Outcome: Late Grade ≥ 3 Gastrointestinal (GI) and Genitourinary (GU) Toxicity of Interest, Using the CTCAE v4.0
Description: Toxicity will be defined as an adverse event possibly, probably, or definitely related to proton beam therapy. A late GI or GU toxicity will be defined as a GI or GU toxicity that occurs between 3 months and 2 years from the completion of proton beam therapy. All patients meeting the eligibility criteria who have signed a consent form and have begun treatment will be evaluable for late toxicity, with the exception of patients determined to be a major violation.
Time Frame: Between 3 months and 24 months post proton beam therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Hypofractionation Proton Beam Therapy
Number analyzed (Participants) | 54
Participants
  GI grade ≥ 3 | 1
  GU grade ≥ 3 | 0

2. Secondary Outcome: Late Grade ≥ 2 GI and GU Toxicity of Interest, Using the CTCAE v4.0
Description: as for outcome 1
Time Frame: Between 3 months and 24 months post proton beam therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Hypofractionation Proton Beam Therapy
Number analyzed (Participants) | 54
Participants
  GI grade ≥ 2 | 6
  GU grade ≥ 2 | 19

3. Secondary Outcome: Acute Grade ≥ 3 GI and GU Toxicity of Interest Within 3 Months Post Proton Beam Therapy, Using the CTCAE v4.0
Description: Toxicity will be defined as an adverse event possibly, probably, or definitely related to proton beam therapy. All patients meeting the eligibility criteria who have signed a consent form and have begun treatment will be evaluable for late toxicity, with the exception of patients determined to be a major violation
Time Frame: Within 3 months post proton beam therapy
Measure: Count of Participants; unit: Participants
Groups:
- Hypofractionation Proton Beam Therapy: Hypofractionation Proton beam therapy with Concurrent Treatment of the Prostate and Pelvic Nodes>
  >>>
  >>
  >>>
  >
  >>>
  >>
  >>> Hypofractionation Proton beam therapy with Concurrent Treatment of the Prostate and Pelvic Nodes
Arm/Group | Hypofractionation Proton Beam Therapy
Number analyzed (Participants) | 55
Participants
  GI grade ≥ 3 | 0
  GU grade ≥ 3 | 0

4. Secondary Outcome: Disease-free Survival Including Freedom From PSA Relapse at 5 Years Post Proton Beam Therapy
Description: Disease-free survival is defined as the time from registration until the time of the first occurrence of biochemical failure, local recurrence, regional recurrence, distant metastases, or death due to any cause. The distribution of disease-free survival will be estimated using the method of Kaplan-Meier.
Time Frame: 5 years post proton beam therapy
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Hypofractionation Proton Beam Therapy
Number analyzed (Participants) | 54
percentage of participants | 90 [81 to 99]

5. Secondary Outcome: Disease-specific Survival at 5 Years Post Proton Beam Therapy
Description: as for outcome 4
Time Frame: 5 years post proton beam therapy
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Hypofractionation Proton Beam Therapy: Hypofractionation Proton beam therapy with Concurrent Treatment of the Prostate and Pelvic Nodes >>>
  >
  >>>
  >>>
  >
  >>> Hypofractionation Proton beam therapy with Concurrent Treatment of the Prostate and Pelvic Nodes
Arm/Group | Hypofractionation Proton Beam Therapy
Number analyzed (Participants) | 54
percentage of participants | 89 [80 to 99]

ADVERSE EVENTS:
Time Frame: 5 years post proton beam therapy
Arm/Group | Hypofractionation Proton Beam Therapy
All-Cause Mortality (participants affected / at risk) | 0/55
Serious Adverse Events (participants affected / at risk) | 0/55
Other Adverse Events (participants affected / at risk) | 55/55
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hypofractionation Proton Beam Therapy (N=55)
Diarrhea (Gastrointestinal disorders) | 25 (89)
Fecal incontinence (Gastrointestinal disorders) | 7 (12)
Proctitis (Gastrointestinal disorders) | 13 (48)
Rectal hemorrhage (Gastrointestinal disorders) | 22 (81)
Rectal stenosis (Gastrointestinal disorders) | 1 (2)
Rectal ulcer (Gastrointestinal disorders) | 1 (2)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2)
Bladder spasm (Renal and urinary disorders) | 2 (5)
Cystitis noninfective (Renal and urinary disorders) | 5 (13)
Hematuria (Renal and urinary disorders) | 8 (11)
Urinary frequency (Renal and urinary disorders) | 55 (607)
Urinary incontinence (Renal and urinary disorders) | 13 (49)
Urinary retention (Renal and urinary disorders) | 40 (233)
Urinary tract obstruction (Renal and urinary disorders) | 33 (201)
Urinary tract pain (Renal and urinary disorders) | 26 (95)
Urinary urgency (Renal and urinary disorders) | 51 (410)
Erectile dysfunction (Reproductive system and breast disorders) | 54 (564)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-10-24): https://cdn.clinicaltrials.gov/large-docs/14/NCT02874014/Prot_SAP_000.pdf
  • Informed Consent Form (2018-07-13): https://cdn.clinicaltrials.gov/large-docs/14/NCT02874014/ICF_001.pdf